CLINICAL TRIAL: NCT00988962
Title: Substance Abuse Treatment for High Risk Chronic Pain Patients on Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Robert N. Jamison, PhD, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007p001732
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Substance Abuse
Keywords: pain; opioids
MeSH Terms: conditions — Substance-Related Disorders; Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-Risk No Treatment (No Intervention)
- High-Risk Treatment (Experimental)
  Interventions: Behavioral: cognitive behavioral training
- Low-Risk (No Intervention)

INTERVENTIONS:
Behavioral: cognitive behavioral training — electronic diaries, compliance checklists, urine screens, individual and group motivational counseling
  Other Names: compliance contract; therapy
  Arms: High-Risk Treatment

SUMMARY:
Chronic back pain patients are often dismissed from a pain center or a primary care practice when they are noncompliant with opioid therapy, instead of being offered treatments to reduce misuse and to improve compliance. Unfortunately, there are few treatment resources for such patients. This study seeks to remedy that problem, with the goal of reducing the rate of prescription opioid misuse among noncompliant patients through the use of novel tracking, education, and counseling interventions.

DETAILED DESCRIPTION:
This study will evaluate drug misuse behavior over 6 months with the use of self-report questionnaires, physician ratings, urine toxicology screens, and electronic diary data.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain for >6 months
* history of taking daily opioids for pain for >6 months
* average >3 on a pain intensity scale of 0 to 10 over past week
* able to speak and understand English
* chronic neck or back pain as primary pain complaint
* willingness to participate

Exclusion Criteria:

* current opioid addiction (M.I.N.I. Section K)
* current diagnosis of cancer or any other malignant disease
* acute osteomyelitis or acute bone disease
* nonambulatory
* present or past DSM-IV diagnosis of schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder
* pregnancy
* any clinically unstable systemic illness judged to interfere with treatment
* an acute condition requiring surgery
* taking opioids intermittently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Drug Misuse Index: 1) physician ratings of misuse (ABC), 2) structured self-report interview (PDUQ), and 3) urine tox screens | All subjects will be followed for 6 months.

SECONDARY OUTCOMES:
1) Rate of patient dismissal from a pain center, 2) treatment satisfaction ratings | Subjects will be followed for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Jamison, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital Pain Management Center, Chestnut Hill, Massachusetts, United States

REFERENCES:
- [Background] Wasan AD, Butler SF, Budman SH, Fernandez K, Weiss RD, Greenfield SF, Jamison RN. Does report of craving opioid medication predict aberrant drug behavior among chronic pain patients? Clin J Pain. 2009 Mar-Apr;25(3):193-8. doi: 10.1097/AJP.0b013e318193a6c4. PMID 19333168
- [Background] Wasan AD, Michna E, Janfaza D, Greenfield S, Teter CJ, Jamison RN. Interpreting urine drug tests: prevalence of morphine metabolism to hydromorphone in chronic pain patients treated with morphine. Pain Med. 2008 Oct;9(7):918-23. doi: 10.1111/j.1526-4637.2007.00354.x. Epub 2007 Aug 28. PMID 18616432
- [Background] Butler SF, Fernandez K, Benoit C, Budman SH, Jamison RN. Validation of the revised Screener and Opioid Assessment for Patients with Pain (SOAPP-R). J Pain. 2008 Apr;9(4):360-72. doi: 10.1016/j.jpain.2007.11.014. Epub 2008 Jan 22. PMID 18203666
- [Background] Marceau LD, Link C, Jamison RN, Carolan S. Electronic diaries as a tool to improve pain management: is there any evidence? Pain Med. 2007 Oct;8 Suppl 3:S101-9. doi: 10.1111/j.1526-4637.2007.00374.x. PMID 17877520
- [Background] Butler SF, Budman SH, Fernandez KC, Houle B, Benoit C, Katz N, Jamison RN. Development and validation of the Current Opioid Misuse Measure. Pain. 2007 Jul;130(1-2):144-56. doi: 10.1016/j.pain.2007.01.014. Epub 2007 May 9. PMID 17493754
- [Background] Akbik H, Butler SF, Budman SH, Fernandez K, Katz NP, Jamison RN. Validation and clinical application of the Screener and Opioid Assessment for Patients with Pain (SOAPP). J Pain Symptom Manage. 2006 Sep;32(3):287-93. doi: 10.1016/j.jpainsymman.2006.03.010. PMID 16939853
- [Background] Butler SF, Budman SH, Fernandez K, Jamison RN. Validation of a screener and opioid assessment measure for patients with chronic pain. Pain. 2004 Nov;112(1-2):65-75. doi: 10.1016/j.pain.2004.07.026. PMID 15494186
- [Background] Michna E, Ross EL, Hynes WL, Nedeljkovic SS, Soumekh S, Janfaza D, Palombi D, Jamison RN. Predicting aberrant drug behavior in patients treated for chronic pain: importance of abuse history. J Pain Symptom Manage. 2004 Sep;28(3):250-8. doi: 10.1016/j.jpainsymman.2004.04.007. PMID 15336337
- [Background] Nedeljkovic SS, Wasan A, Jamison RN. Assessment of efficacy of long-term opioid therapy in pain patients with substance abuse potential. Clin J Pain. 2002 Jul-Aug;18(4 Suppl):S39-51. doi: 10.1097/00002508-200207001-00005. PMID 12479253